CLINICAL TRIAL: NCT06391060
Title: Gender Differences in Robotic Surgery for Rectal Cancer: a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Daorong Wang (Other)
Responsible Party: Sponsor-Investigator, Daorong Wang, Professor, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Other Study IDs: ali005
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Rectal Cancer; Gender; Complication,Postoperative; Surgery-Complications
MeSH Terms: conditions — Rectal Neoplasms; Coitus; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient characteristics group: Retrospective evaluation and comparison of demographic characteristics, pre-operative TNM stage, distance from anal verge, tumor size, tumor grade, American Society of Anesthesiologists (ASA) score, and body mass index (BMI) were conducted among both patient groups. Peri-operative and post-operative data, including morbidity and mortality, were assessed, alongside parameters such as distal resection margin (DRM), proximal resection margin (PRM), harvested lymph nodes (HLN), and Clavien-Dindo Classification (CDC) scores. Diagnosis of anastomotic leakage was confirmed by clinical suspicion (e.g., changes in drainage, fever, abdominal pain) and further validated through contrast enema observed during follow-up computed tomography (CT). Hospital stay and readmission rates were monitored for up to 90 days post-surgery.
  Interventions: Procedure: Impact of Gender on Davinci rectal surgery
- Post-operative group: Post-operative outcomes encompassed operative duration, estimated blood loss, time to first flatus passage, duration of liquid diet, and length of hospital stay following surgery. Operative duration comprised the time from initial skin incision to closure, including the time needed for robotic surgery docking and undocking. Upon experiencing initial flatulence, patients transitioned to a liquid diet. Hospital stay duration was measured from the time of surgery to discharge. The overall cost of surgery, including surgical procedures, anesthesia, medications, and post-operative care, was considered in the total expenditure analysis
  Interventions: Procedure: Impact of Gender on Davinci rectal surgery

INTERVENTIONS:
Procedure: Impact of Gender on Davinci rectal surgery — gender-specific considerations in the surgical management and post-operative care of rectal cancer patients undergoing robotic surgery
  Other Names: Davinci

SUMMARY:
Objective: To investigate gender-based differences in outcomes following robotic surgery for rectal cancer.

Methods: A retrospective study was conducted on 155 patients (82 males, 73 females) who underwent robotic surgery for rectal cancer. Demographic, pre-operative, operative, and post-operative data were collected and analyzed.

Pre-operative study:

All patients underwent a standardized pre-operative work-up, which included a physical examination, comprehensive colonoscopy with biopsy, rigid rectoscopy, pelvic magnetic resonance imaging (MRI) scan, computed tomography (CT) of the thorax and abdomen, and measurement of carcinoembryonic antigen (CEA) levels. Tumor staging followed the TNM staging criteria (American Joint Committee on Cancer), with the T and N stages determined by the most advanced findings from any imaging modality

Data collected:

Retrospective evaluation and comparison of demographic characteristics, pre-operative TNM stage, distance from anal verge, tumor size, tumor grade, American Society of Anesthesiologists (ASA) score, and body mass index (BMI) were conducted among both patient groups. Peri-operative and post-operative data, including morbidity and mortality, were assessed, alongside parameters such as distal resection margin (DRM), proximal resection margin (PRM), harvested lymph nodes (HLN), and Clavien-Dindo Classification (CDC) scores. Diagnosis of anastomotic leakage was confirmed by clinical suspicion (e.g., changes in drainage, fever, abdominal pain) and further validated through contrast enema observed during follow-up computed tomography (CT). Hospital stay and readmission rates were monitored for up to 90 days post-surgery.

Post-operative follow-up:

Post-operative outcomes encompassed operative duration, estimated blood loss, time to first flatus passage, duration of liquid diet, and length of hospital stay following surgery. Operative duration comprised the time from initial skin incision to closure, including the time needed for robotic surgery docking and undocking. Upon experiencing initial flatulence, patients transitioned to a liquid diet. Hospital stay duration was measured from the time of surgery to discharge. The overall cost of surgery, including surgical procedures, anesthesia, medications, and post-operative care, was considered in the total expenditure analysis.

ELIGIBILITY:
Inclusion Criteria:

A confirmed histological diagnosis of colorectal malignancy was a prerequisite for enrollment in this study. Additionally, obtaining informed consent from patients for surgical intervention was mandatory.

Exclusion Criteria:

Patients with bleeding of the gastrointestinal tract, inflammatory bowel disease, synchronous tumors, benign conditions, and clinical T4 stage tumors unresponsive to neoadjuvant therapy were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Our institution, a government-affiliated university hospital, conducts various robotic procedures encompassing colorectal, hepato-biliary, gastro-esophageal, and retro-peritoneal surgeries. A comprehensive database of laparoscopic and robotic rectal surgeries has been established, with prospective data collection spanning from July 2021 to March 2024. Approval for the study was obtained from the institutional review board at Northern Jiangsu People's Hospital, and all operations were conducted utilizing the da Vinci Robotic Surgical System model Xi, manufactured by Intuitive Surgical, located in Sunnyvale, CA, USA.
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Gender Differences in Robotic Surgery for Rectal Cancer: a retrospective study | 15th of April 2024
  gender-specific considerations in the surgical management and post-operative care of rectal cancer patients undergoing robotic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China